CLINICAL TRIAL: NCT06398431
Title: A Study on Validation of Gait Analysis Wireless Small Inertial Sensor and Diagnostic Machine Learning Model for Classification of Elderly Fall Risk Group
Brief Title: Validating Wireless Gait Sensor for Elderly Fall Risk Classification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Collaborators: Pusan National University (Other)
Responsible Party: Principal Investigator, Sungchul Huh, Assistant Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-2023-001
Record Dates: First submitted 2023-12-21; First posted 2024-05-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Elderly Person
Keywords: Fall Risk Assessment; Walking analysis; Machine Running

STUDY DESIGN:
Intervention Model Description: The subject wears shoes equipped with sensors, and walks for 1 minute, repeating this three times. We plan to machine learn the correlation between walking data and BBS data. Since machine learning becomes more accurate as the number increases, the analysis group was set at 51 people.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait group (Experimental): 1. Those aged 55 years or older
  2. Those who can walk independently for at least 1 minute
  3. Those who are not taking medications that affect the ability to maintain balance
  4. Those who have not had any orthopedic problems such as lower limb fractures within the past 6 months
  Interventions: Device: Walking analysis sensor

INTERVENTIONS:
Device: Walking analysis sensor — Participant gait analysis with the inertial sensor

SUMMARY:
The walking status of elderly patients over 65 years of age in the hospital will be verified through political analysis and objective fall risk assessment through wireless inertial sensors and diagnostic machine learning models, and based on the results, As investigators, providing a foundation for the objective evaluation of the risk of falling patients by nurses in general wards in the future.

DETAILED DESCRIPTION:
Currently, in the case of general clinical wards in Korea, the evaluator who assesses the risk of falling during the patient's hospitalization changes every time, and the evaluation of fall risk differs for the same patient depending on the subjectivity of the evaluator. Hence, evaluating falls requires assessing the patient's walking based on consistent criteria. Through walking analysis with a wireless small inertial sensor, there is an expectation that the incidence of fall risk will decrease. When analyzing walking to classify fall risk groups, quantitative evaluation should be applied for stride length, gait speed, step width, cadence, and gait cycle, but currently, fall assessments taking this into account are not properly conducted. Therefore, it is necessary to prepare and apply quantitative standards for fall evaluation through walking analysis through wireless small inertial sensors and data machine learning to classify the risk of falling in elderly hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

1. a person over the age of 55
2. Persons who can walk independently for at least one minute
3. Those who do not take drugs that affect their ability to maintain balance
4. A person who does not have an orthopedic problem such as a fracture of the lower extremities within six months

Exclusion Criteria:

1. Those who have difficulty understanding the gait analysis program or difficulty expressing symptoms
2. A person deemed unfit for this study by a rehabilitation specialist due to other conditions
3. A person who is unable to apply this walking analysis program due to serious cardiovascular diseases

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Falls Risk Assessment Scale | Patient gait data is collected continuously throughout the study period, enabling the ongoing measurement of falls risk.
  A falls risk assessment scale measured through the analysis of patients' gait using wireless inertial sensors and a diagnostic machine learning model.

CONTACTS AND LOCATIONS:
Overall Officials: Sungchul Huh, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Sungchul Huh, MD, Yangsan, South Korea